CLINICAL TRIAL: NCT02019173
Title: Rehabilitation Boot Camp: an Innovative, Four-Week Program to Deliver Intensive Balance and Mobility Therapy to People With Acquired Brain Injury (ABI)
Brief Title: Rehabilitation Boot Camp: Intensive Balance and Mobility Therapy for People With Acquired Brain Injury
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Manitoba (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: H2013:403
Record Dates: First submitted 2013-12-09; First posted 2013-12-24 (Estimated); Last update posted 2015-03-24 (Estimated); Status verified 2013-12

CONDITIONS: Brain Injuries
Keywords: exercise therapy; brain injury; postural balance
MeSH Terms: conditions — Brain Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Boot camp balance training (Experimental): Intense physical rehabilitation directed at improving balance and mobility will be provided to individuals in a group setting (6 participants in a group) for 4 weeks, 3 days a week for 6 hours per day.
  Interventions: Behavioral: Boot Camp Balance Training

INTERVENTIONS:
Behavioral: Boot Camp Balance Training — Intense physical rehabilitation directed at improving balance and mobility will be provided to individuals in a group setting (6 participants in a group) for 4 weeks, 3 days a week for 6 hours per day.

SUMMARY:
The purpose of this study is to determine

1. if it is practical to treat moderately to severely brain injured patients who have problems with their balance and mobility in a group "boot camp" (3 days a week, 6 hours/day for 4 weeks) exercise class.
2. If they show improvements compared to 4 weeks of not receiving this treatment
3. If electronic daily monitoring of their center of foot pressure during a standardized balance task will allow us to see small changes in ability.

A baseline assessment of all outcome measures will be performed. This will be repeated 4 weeks later. The intervention will be delivered (4 weeks) and a follow up assessment of all outcome measures will be performed one week later. A follow up of the Primary outcome measure, the PART-O participation questionnaire will be done 12 weeks later.

Participants will attend group therapy consisting of a variety of exercises designed specifically to target balance and mobility deficits and based on the concept that through Repetitive Functional Task Practice (RFTP), recovery of function can occur as the result of neural adaptation. Exercises will be both individualized (delivered in a circuit) and group activities. Supervision and guidance will be provided by a registered Physical Therapist and a Rehabilitation Assistant. During the intervention, the amount and type of RFTP, any adverse events, and any need for extra staff will be recorded on a daily basis. As well, a standardized individualized task will be performed with center of foot pressure recording on a daily basis.

Analysis: changes in outcome measures immediately after the non-intervention compared to the after the intervention period will be statistically determined to estimate efficacy of this treatment model. Descriptive measures of RFTP time/day, staffing levels/day and adverse events will be used to support feasibility and safety of this model.

DETAILED DESCRIPTION:
See below for details about outcome measures and eligibility criteria.

ELIGIBILITY:
Inclusion Criteria:

* Moderate to Severe Acquired Brain Injury due to trauma, anoxia or infection, one to five years since onset
* Re: Physical Function:

  * Able to sit independently unsupported at the edge of the bed
  * Able to assist rising from sit to stand
  * Able to stand unsupported (with or without supervision) for at least thirty seconds.
  * Standing tolerance of at least 3 minutes (may use upper limb support to stabilize).
  * Able to voluntarily move at least one leg (with or without synergic movements).
  * Functional use of at least one arm and able to lift to 90˚ shoulder elevation.
  * If the person is able to walk independently, he or she requires a walking aide, has difficulty walking outdoors or on uneven terrain, and/or demonstrates an abnormal gait pattern.
  * Medically stable and with the tolerance to be physically and mentally active over the treatment day with appropriate rests.
  * Can safely and independently eat, drink and use a toilet OR availability of an assistant to help with these functions.
* Sufficient Cognitive ability to provide informed consent.
* English communication at a level to understand instruction and provide informed consent.
* Impulse control and social skills to allow group participation with only occasional redirection from therapy staff

Exclusion Criteria:

* ABI due to primary Cerebral Vascular Accident (Stroke).
* Mild ABI/concussion.
* not able to perform the above physical criteria, OR regularly walking in all conditions, outdoors without a walking aide and without any apparent gait deficit will not be eligible.
* Unwilling to provide permission for researchers to obtain medical approval to participate in program.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 12 (Estimated)
Dates: Start 2014-06; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Change from baseline measure of Dual Task Cost of a visual cognitive task on stationery balance | This will be assessed 5 weeks prior, 1 week prior, 1 week post intervention
  The sway path length (SPL) will be recorded while standing unsupported. The performance on a visual spatial task will be recorded using a computer program that is based on the Useful Field of View test while the subject is in supported sitting. Then the balance task and cognitive task will be performed simultaneously to generate a Dual Task Cost in performance.

SECONDARY OUTCOMES:
Change from baseline measure in time (seconds) to perform Five Times Sit to Stand Test | 5 weeks, 1 week prior and 1 week post intervention
Change in score from baseline measure in Chedoke McMaster Stroke Assessment Activity Scale | 5 weeks, 1 week prior and 1 week post intervention
  A variety of functional mobility tasks including bed mobility, transfers, walking and stairs are performed and rated on a 7-point scale
Change from baseline measure of the Sway Path Length during The Modified Clinical Test of Integration in Balance (mCTSIB) | 5 weeks, 1 week prior and 1 week post intervention
  Ability to maintain still standing is assessed in 4 sensory conditions; on a solid surface eyes open, on a sponge surface eyes open, on a solid surface eyes closed and on a sponge surface eyes closed
Change in distance walked (meters) from baseline measure in the Two Minute Walk Test (2 MWT) | 5 weeks, 1 week pre and 1 week post intervention.
Change in score from baseline measure in the Participation Assessment with Recombined Tools - Objective 17 (PART-O 17) | This will be performed at the following time points: 5 weeks prior to the intervention, 1 week prior to the intervention, one week after the intervention and 12 weeks after the intervention
  This is an interview-style questionnaire to quantify subject participation in the following domains; productivity, social relations and "out and about". It has been specifically developed for the brain injured population.

OTHER OUTCOMES:
Number of Adverse Events | This will be recorded on a daily basis on days that participant is receiving the intervention
  Any change in health status will b recorded and categorized into either not related to intervention or related to the intervention. Those that are related to the intervention will be further categorized into "anticipated", "unanticipated minor" (i.e not requiring medical attention) and "unanticipated major"(requiring medical attention).
Level of staffing required | This will be recorded on a daily basis on the days that participants receive the intervention (4 weeks)
  For every participant attendance day the number of therapy staff members required will be recorded.
Amount and of Function Repetitive Task Practice per Treatment Day | This will be recorded on a daily basis on the days that participants receive the intervention (4 weeks)
  The duration of all planned therapy activities will be recorded on each participant treatment day, to allow an average for each activity to be generated
Change from baseline on Balance Performance during an Individualized Task from ba | 5 weeks, 1 week, every treatment day during the intervention, and 1 week post intervention
  Center of foot pressure (COP) measures will be taken during an individualized rhythmic balance task, selected on the basis of the participants needs and level of ability. This will allow within-subject analysis to determine trajectory of balance skill change.

CONTACTS AND LOCATIONS:
Overall Officials: Cristabel Nett, BMR(PT), Principal Investigator — University of Manitoba (MSc candidate)
Locations (1):
- University of Manitoba, School of Medical Rehabilitation, Winnipeg, Manitoba, Canada